CLINICAL TRIAL: NCT06441838
Title: The Effect of Listening to the Inshirah Surah on Depression, Anxiety, Stress and Mental Well-Being in Hemodialysis Patients.
Brief Title: The Effect of Listening to Surah Inshirah on Mental Health in Hemodialysis Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Omer Tanriverdi, Asistant Professor, Mardin Artuklu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Mardin Artuklu Üniversitesi
Record Dates: First submitted 2024-04-20; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Hemodialysis Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Listening to Surah Inshirah (Experimental): Experimental group patients; A patient descriptive characteristics form will be administered, and the pre-test Depression, Stress, Anxiety Scale and Warwick-Edinburgh Mental Well-Being Scale will be administered. Then, Surah Inshirah will be listened to and the final test, Depression, Stress, Anxiety Scale and Warwick-Edinburgh Mental Well-Being Scale will be administered.
  Interventions: Behavioral: Surah Inshirah
- control group (No Intervention): intervention group patients; Patient descriptive characteristics form, Depression, Stress, Anxiety Scale and Warwick-Edinburgh Mental Well-Being Scale will be administered. Then, the Depression, Stress, Anxiety Scale and Warwick-Edinburgh Mental Well-Being Scale will be administered 1 month later without any intervention.

INTERVENTIONS:
Behavioral: Surah Inshirah — The effects of Surah Al-Inshirah on patients' depression, anxiety, stress and mental well-being will be evaluated during hemodialysis in the experimental group.
  Arms: Listening to Surah Inshirah

SUMMARY:
In addition to physical symptoms, mental, social and economic problems may also occur in patients receiving hemodialysis treatment. The most prominent among these problems are psychological problems. It is known that depression and anxiety levels are high in hemodialysis patients.Non-pharmacological methods reduce the patient's pain and anxiety by creating a feeling of comfort and control in the patient. Relaxation techniques such as hypnosis, yoga and music are among these. The main purpose of these methods is to draw the attention of the individual in another direction. Praying is also one of the non-drug methods, and the number of studies on this subject is very limited, and there are studies where it has been determined that praying and praying reduces the anxiety levels of patients.Purpose: To examine the effect of listening to Surah Inshirah on depression, anxiety, stress and mental well-being of hemodialysis patients during treatment.

Method: The population of the research will consist of hemodialysis patients who are treated at Mardin Training and Research Hospital, meet the inclusion criteria and volunteer to participate in the research.

The study group of 60 people who will participate in the research will be divided into two equal groups according to the table of random numbers obtained from the computer-based Research Randomizer program.

Experimental group patients; A patient descriptive characteristics form will be applied, and the pre-test depression, anxiety, stress and mental well-being scale will be applied. Then, Surah Inshirah will be listened to and the final test, the depression, anxiety, stress and mental well-being scale, will be applied.

Control group patients; A patient descriptive characteristics form will be applied, and the depression, anxiety, stress and mental well-being scale will be applied. The final test will be applied to the depression, anxiety, stress and mental well-being scale without any intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can be contacted,Patients aged 18 and over were included in the study.

Exclusion Criteria:

* Patients aged 18 and over were included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-03-23 (Actual); Study Completion 2024-03-23 (Actual)

PRIMARY OUTCOMES:
patient information form | Baseline (It will be applied to patients before hemodialysis)
  This form, created by the researcher with the support of the relevant literature, consists of 8 questions that question the patients' education level, age, gender, profession, marital status, income level, with whom they live, and duration of illness.

SECONDARY OUTCOMES:
depression anxiety stress scale | Baseline (It will be applied to patients before hemodialysis)
  It consists of 7 depression, 7 anxiety and 7 stress questions.

OTHER OUTCOMES:
mental well-being scale | Baseline (It will be applied to patients before hemodialysis)
  It consists of 14 questions

CONTACTS AND LOCATIONS:
Locations (1):
- Ömer TANRIVERDİ, Mardin, Turkey (Türkiye)